CLINICAL TRIAL: NCT00894881
Title: The Effect of Colonoscopy on Resting Energy Expenditure
Status: Unknown | Type: Observational
Last Known Status: Not yet recruiting
Sponsor: Tel-Aviv Sourasky Medical Center (Other Government)
Responsible Party: Prof' Nachum Vaisman, Tel-Aviv Sourasky Medical Center
Other Study IDs: TASMC-09-NV-0080-CTIL
Record Dates: First submitted 2009-05-06; First posted 2009-05-07 (Estimated); Last update posted 2009-05-07 (Estimated); Status verified 2009-05

CONDITIONS: Healthy
Keywords: colonoscopy; Healthy individuals before colonoscopy

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No

GROUPS / COHORTS (1):
- 1 group: patients before colonoscopy
  Interventions: Procedure: Gut cleaning as a preparation to colonoscopy [resting energy expenditure (REE)]

INTERVENTIONS:
Procedure: Gut cleaning as a preparation to colonoscopy [resting energy expenditure (REE)] — resting energy expenditure (REE).
  Other Names: resting energy expenditure (REE).

SUMMARY:
The Effect of Gut Cleaning as a Preparation to Colonoscopy on resting energy expenditure (REE).

ELIGIBILITY:
Inclusion Criteria:

* Healthy individuals before colonoscopy

Exclusion Criteria:

* None

Min Age: 18 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Study Population: Healthy individuals before colonoscopy
Sampling Method: Non-Probability Sample
Enrollment: 30 (Estimated)
Dates: Start 2009-05; Primary Completion 2010-05 (Estimated); Study Completion 2010-05 (Estimated)

PRIMARY OUTCOMES:
To measure the Effect of Gut Cleaning as a Preparation to Colonoscopy on resting energy expenditure (REE). | 1 year

CONTACTS AND LOCATIONS:
Overall Officials: Nachum Vaisman, Prof', Principal Investigator — Tel-Aviv Sourasky Medical Center
Locations (1):
- Tel-Aviv Sourasky Medical Center, Tel Aviv, Israel